CLINICAL TRIAL: NCT07367737
Title: Histatin-1 Levels in Smokers and Non-smokers With Periodontitis Patients: A Comparative Study Before and After Nonsurgical Periodontal Therapy (Prospective Clinical Trial)
Brief Title: Histatin-1 Levels in Smokers and Non-smokers With Periodontitis Patients: A Comparative Study Before and After Nonsurgical Periodontal Therapy
Acronym: NSPT
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Aqeel Ali, Assistant lecturer, University of Baghdad
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: UBaghdad
Record Dates: First submitted 2025-11-23; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-12

CONDITIONS: Periodontitis; Periodontal Diseases
Keywords: periodontitis, NSPT
MeSH Terms: conditions — Periodontitis; Periodontal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- smokers periodontitis (Other): 25 smokers with probing depth (4-6mm), unstable periodontitis were enrolled in the study and underwent NSPT. Saliva samples were obtained prior to, and one month and three months subsequent to, NSPT. By employing an enzyme-linked immunosorbent assay (ELISA)
  Interventions: Procedure: Non Surgical Periodontal Treatment
- non smokers periodontitis (Other): 25 non smokers with probing depth (4-6mm), unstable periodontitis were enrolled in the study and underwent NSPT. Saliva samples were obtained prior to, and one month and three months subsequent to, NSPT. By employing an enzyme-linked immunosorbent assay (ELISA)
  Interventions: Procedure: Non Surgical Periodontal Treatment

INTERVENTIONS:
Procedure: Non Surgical Periodontal Treatment — All patients underwent clinical evaluation and were provided with oral hygiene instructions followed by supragingival full-mouth scaling with an ultrasonic scaler (WOODPECKER® UDS-K). They were also told to use dental floss and interdental brushes on need and to brush their teeth twice a day. The examiner provided each patient with a toothbrush and toothpaste. The subjects were scheduled to undergo non-surgical periodontal treatment of the clinic one week after the previous appointment, that included instructions on oral hygiene and periodontal treatment with root debridement with Gracey curette
  Arms: non smokers periodontitis
Procedure: Non Surgical Periodontal Treatment — All patients underwent clinical evaluation and were provided with oral hygiene instructions followed by supragingival full-mouth scaling with an ultrasonic scaler (WOODPECKER® UDS-K). They were also told to use dental floss and interdental brushes on need and to brush their teeth twice a day. The examiner provided each patient with a toothbrush and toothpaste. The subjects were scheduled to undergo non-surgical periodontal treatment of the clinic one week after the previous appointment, that included instructions on oral hygiene and periodontal treatment with root debridement with Gracey curette.
  Arms: smokers periodontitis

SUMMARY:
This study evaluated the impact of smoking on salivary histatin-1 levels and clinical healing in 50 patients with unstable periodontitis (25 smokers and 25 non-smokers) undergoing non-surgical periodontal therapy (NSPT). By measuring clinical parameters like probing depth and clinical attachment level alongside ELISA-based protein analysis at baseline, one month, and three months post-treatment, the researchers sought to determine if the impaired wound healing typically seen in smokers correlates with a suppressed expression of this specific salivary protein.

DETAILED DESCRIPTION:
Periodontal disease is a chronic progressive destructive disease of the tissues supporting the teeth, collectively known as the periodontium. The main clinical parameters of periodontal diseases are clinical attachment loss , radiographic reduced alveolar bone height, probing depth and bleeding on probing. If untreated, teeth can be lost, but most cases can be prevented and treated . In recent definitions of periodontitis, smoking is considered the most important environmental risk factor. . Furthermore, The severity of periodontitis is directly influenced by the smoking habits of an individual and the number of cigarettes smoked per day. Smoking increases the risk of periodontitis , by compromising the host's immune response, thereby reducing the ability to combat periodontal pathogens. Additionally, it impairs the circulation of blood to periodontal tissues, which hinders healing processes and fosters an environment conducive to bacterial proliferation. These factors collectively contribute to enhanced inflammation, periodontal tissue destruction, and the accelerated progression of periodontal disease.

In general, Histatin, a group of histidine-rich proteins, exhibit diverse functions, including antifungal, bactericidal, and enamel-protective activities. Histatin-1 is a naturally occurring antimicrobial peptide found in human saliva, known for its role in oral health and immunity. It has garnered significant attention in the context of periodontal disease due to its multifaceted biological functions. Histatin-1 demonstrates significant antibacterial efficacy against many oral infections, involving bacteria, fungi, and viruses. In periodontal disease, pathogenic bacteria such as Porphyromonas gingivalis, Tannerella forsythia, and Treponema denticola play a critical role in disease progression. Histatin-1 disrupts the cell membranes of these pathogens, leading to their destruction and helping to maintain microbial balance in the oral cavity.

Histatin-1 has been shown to modulate inflammatory responses by inhibiting the production of pro-inflammatory cytokines, such as IL-6, IL-8, and TNF-α. Therefore, reducing tissue damage and promotes healing in periodontal tissues6. Histatin-1 plays a significant role in promoting the migration and proliferation of epithelial cells, which is crucial for the regeneration of periodontal tissues. It accelerates wound closure and tissue repair, making it a potential therapeutic agent for managing periodontal lesions and promoting periodontal regeneration.

Biofilm formation by pathogenic bacteria is a crucial determinant in the onset and progression of periodontal disease. Histatin-1 has been found to inhibit biofilm formation by interfering with bacterial adhesion and aggregation, this property helps prevent the colonization of pathogenic bacteria on tooth surfaces and periodontal tissues. Histatin-1 interacts with host immune cells, such as neutrophils and macrophages, enhancing their ability to combat infections. It also modulates the immune response to prevent excessive inflammation, which can lead to tissue destruction in periodontal disease. Furthermore, research has broadened the range of cell types responsive to histatin-1, demonstrating its capacity to stimulate osteogenic differentiation and facilitate mineralization in pre-osteoblasts, as well as mesenchymal cells sourced from tooth pulp and apical papilla. These findings offer fresh perspectives on the physiological significance of histatin-1's effects across diverse cell populations within the oral cavity. Given its antimicrobial, anti-inflammatory, and wound-healing properties, Histatin-1 is being explored as a potential therapeutic agent for periodontal disease. It could be incorporated into mouthwashes, gels, or local drug delivery systems to target periodontal pockets and promote oral health Non-surgical periodontal approach, including scaling and root surface debridement (RSD) as well as oral hygiene instructions, is the most effective treatment for periodontitis . The goal of the treatment is to eliminate the biofilm that has built up on the teeth surfaces ., supra and subgingival, and delay the recolonization of the sites by periodontopathogens. Studies indicate that these treatments can halt the progression of periodontitis in pockets ranging from shallow to moderate. Salivary biomarkers serve as valuable diagnostic and prognostic indicators for periodontal disease, as well as markers for monitoring the healing process .

ELIGIBILITY:
Inclusion Criteria:

* the present study required participants to be systemically healthy, with no history of systemic diseases such as diabetes mellitus, cardiovascular disease, or renal disease.
* Participants had not undergone periodontal treatment in the past six months or taken any medication in the last three months.
* They also needed to have at least 20 teeth and be diagnosed with moderate periodontitis, characterized by a PPD of 4-6 mm, generalized, unstable periodontitis.

Exclusion Criteria:

* the presence of intraoral plaque-retentive factors such as crowns, bridges, partial dentures, orthodontic appliances, furcation-involved teeth, overhanging restorations, and tooth anomalies.
* Patients who had received antibiotic therapy within the previous three months.

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-01-29 (Estimated); Study Completion 2026-02-10 (Estimated)

PRIMARY OUTCOMES:
Measuring the level of salivary histatin-1 in nonsmoker and smoker patients with unstable periodontitis over the periods of one month, and three months following NSPT | baseline,1 month, 3 months
  Before the clinical examination, 1 mL of unstimulated saliva was collected from every participant in the morning appointment using the drooling method by Navazesh . Patients were asked to remain fasting for 30 min. Saliva was collected via 30-mm diameter round-bottom polypropylene tubes (50-ml Falcon® tubes). Then, 1 ml of saliva was transferred into a 1.5 ml Eppendorf tube contained 10 μl of 2× protease inhibitor (Sigma-Aldrich, St. Louis, MO, USA). The samples were subsequently centrifuged for 5 minutes at 3000 rpm, and the supernatant was frozen at -70 °C for subsequent analyses.

CONTACTS AND LOCATIONS:
Locations (1):
- university of Baghdad, college of dentistry, Baghdad, Medical City, Iraq

IPD SHARING:
Plan to Share IPD: Yes
to disseminate the research idea
Supporting Information: Study Protocol
Time Frame: from 1/5/2025 to 1/12/2025